CLINICAL TRIAL: NCT01970059
Title: Efficacy and Safety Comparison of Extended-Release Carvedilol Sulfate and Sustained-release Metoprolol Succinate in Patients With Hypertension
Brief Title: A Phase Ⅲ Study of Extended-Release Carvedilol Sulfate for the Treatment of Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KWDLEH2012
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended-Release Carvedilol Sulfate (Experimental): 18-72mg/d,po
  Interventions: Drug: Extended-Release Carvedilol Sulfate
- Sustained-release Metoprolol Succinate (Active Comparator): 47.5-190mg/d,po
  Interventions: Drug: Sustained-release Metoprolol Succinate

INTERVENTIONS:
Drug: Extended-Release Carvedilol Sulfate
  Arms: Extended-Release Carvedilol Sulfate
Drug: Sustained-release Metoprolol Succinate
  Arms: Sustained-release Metoprolol Succinate

SUMMARY:
The aim of present study is to evaluate the efficacy and safety of Extended-Release Carvedilol Sulfate versus in Patients With Mild or Moderate Primary Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* Aged from 18 to 70 years
* Had a history of essential hypertension
* Average sitting diastolic blood pressure≧90mmHg，but≦109mmHg

Exclusion Criteria:

* Malignant hypertension
* Average sitting systolic blood pressure≧180mmHg
* Type 2 diabetes with hemoglobin A1c≥9%
* Type 1 diabetes
* New York Heart Association class Ⅱ-Ⅳ congestive heart-failure
* Unstable angina
* Second or third degree heart block or history of sick sinus syndrome unless a pacemaker was in place
* Atrial fibrillation
* Bradycardia (<60 bpm, seated)
* Asthma or other obstructive pulmonary disease
* History of myocardial infarction
* Stroke in the 6 months before screening
* Known contraindications to β-adrenergic blocker therapy
* Glutamic-oxaloacetic transaminase and/or glutamic-pyruvic transaminase>3 times upper limit of normal
* Crea>2 times upper limit of normal
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Sitting Diastolic Blood Pressure (sDBP) at Week 8 | Baseline and Week 8

SECONDARY OUTCOMES:
Mean Change From Baseline in Sitting Systolic Blood Pressure (sSBP) at Week 8 | Baseline and Week 8
Proportion of Patients With Sitting Systolic Blood Pressure <140 mm Hg and Sitting Diastolic Blood Pressure <90 mm Hg at Week 8 | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Yun Zhang, Professor, Principal Investigator — Qilu Hospital of Shandong University
Locations (11):
- China (11):
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Taizhou Hospital, Taizhou, Zhejiang
  - Xuan Wu hospital affiliated to Capital Medical University, Beijing
  - Beijing Tongren hospital affiliated to Capital Medical University, Beijing
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai